CLINICAL TRIAL: NCT03747627
Title: British Pigeon Fanciers Genetics of Interstitial Lung Disease Study
Brief Title: BPF Genetics of ILD Study
Acronym: BPF GILD
Status: Active, not recruiting | Type: Observational
Sponsor: University of Dundee (Other)
Collaborators: University of Leicester (Other); University of Glasgow (Other); Newcastle University (Other); British Lung Foundation (Other); British Pigeon Fanciers Medical Research (Unknown)
Responsible Party: Principal Investigator, Mark Spears, Dr Mark Spears, Consultant in Respiratory Medicine, University of Dundee
Other Study IDs: MS001
Record Dates: First submitted 2018-11-14; First posted 2018-11-20 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Lung; Disease, Interstitial, With Fibrosis; Alveolitis, Extrinsic Allergic; Bird Fancier's Lung; Idiopathic Interstitial Pneumonias; Lung Diseases, Interstitial; Idiopathic Pulmonary Fibrosis
Keywords: Interstitial Lung Disease (ILD); Hypersensitivity Pneumonitis; Idiopathic Pulmonary Fibrosis (IPF); Extrinsic Allergic Alveolitis (EAA); Bird Fancier's Lung; Genetics
MeSH Terms: conditions — Disease; Alveolitis, Extrinsic Allergic; Bird Fancier's Lung; Idiopathic Interstitial Pneumonias; Lung Diseases, Interstitial; Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Blood samples will be prepared for DNA analysis
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: Genetic profiling — All participating subjects will undergo detailed genetic analysis, with the aim of detecting novel genetic drivers for the development of interstitial lung disease in the context of known sensitising agent (pigeon antigen)

SUMMARY:
The investigators aim to examine the genetic determinants of interstitial lung disease in a cohort of subjects with regular exposure to pigeons, a known cause of one form of interstitial lung disease known as hypersensitivity pneumonitis. In addition we will examine immunological causes for hypersensitivity pneumonitis in this group.

We anticipate our work will provide insights of use to clinicians and patients with hypersensitivity pneumonitis and other interstitial lung diseases.

DETAILED DESCRIPTION:
The investigators aim to recruit participants with regular racing pigeon exposure at national (UK) and regional pigeon fancier meetings.

Consenting subjects will complete questionnaires, provide blood samples for genetic analysis and immunological testing and undertake lung function measurements.

Subjects will be observed, and encouraged to report referral to specialist respiratory services, and following this information will be sought on diagnosis (including supporting evidence). Where interstitial lung disease is detected this will be linked to subsequent unbiased analysis to detect potential predisposing genetic associations.

ELIGIBILITY:
Inclusion Criteria:

* regular exposure to racing pigeons

Exclusion Criteria:

* Unwilling to participate

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants in the sport of Pigeon racing
Sampling Method: Non-Probability Sample
Enrollment: 475 (Actual)
Dates: Start 2019-01-19 (Actual); Primary Completion 2025-01-19 (Actual); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Relationship of specific genetic markers to development of interstitial lung disease | 5 years
  Participants will be screened for MUC5B genetic profile to allow examination of MUC5B genetic profile relationship with risk of developing interstitial lung disease in this group

CONTACTS AND LOCATIONS:
Overall Officials: Mark Spears, PhD, FRCP, Principal Investigator — NHS Tayside & University of Dundee; Louise Wain, PhD, Principal Investigator — University of Leicester
Locations (2):
- United Kingdom (2):
  - Scottish Homing Union, Lanark, Lanark
  - Royal Pigeon Racing Association Meeting, Blackpool

IPD SHARING:
Plan to Share IPD: Undecided
Will be considered, dependent on potential for increased power